CLINICAL TRIAL: NCT03260270
Title: Detection of Asymptomatic Venous Thrombosis in Gynecological Patients With Pelvic Masses
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Kero Wagdy, principal investigator, Assiut University
Other Study IDs: ASU
Record Dates: First submitted 2017-08-22; First posted 2017-08-24 (Actual); Last update posted 2017-08-24 (Actual); Status verified 2017-08

CONDITIONS: Silent; Thrombosis
MeSH Terms: conditions — Thrombosis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Week
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: color doppler ultrasound — All patients are going to be examined by color Doppler ultrasound and the high risk patients are going to be examined by direct MDCT venography .
  Other Names: direct MDCT venography

SUMMARY:
Venous thromboembolism (VTE) is a serious preventable complication of gynecological surgery. High incidence of silent VTE before surgery seems attributable to the high incidence of VTE after surgery in ovarian cancer .so the aim of work is to detect silent venous thrombosis in gynecological patients suffering from pelvic masses using different imaging modalities .

DETAILED DESCRIPTION:
High incidence of silent VTE before surgery seems attributable to the high incidence of VTE after surgery in ovarian cancer .

The incidence rate of DVT is about 10% to 40% in medical or general surgical patients without prophylaxis .With prophylaxis, the postoperative incidence of VTE was 1.14% in women with gynecological disease, and 0.7% in patients undergoing laparoscopic gynecological surgery, 0.3% in patients undergoing urogynecological surgery, and 4% in gynecological cancer patients, respectively. Most of published studies enrolled only symptomatic patients with DVT, whereas asymptomatic patients could be easily neglected under the absence of effective detection. In fact, approximately 50% of DVT patients are silent, so the actual incidence of postoperative DVT might be higher than reported . The asymptomatic DVT has been confirmed to increase the development of post-thrombotic syndrome (PTS).

The essence of any surveillance strategy would be the identification of DVT in the expectation that anticoagulation at the presymptomatic stage would prevent fatal pulmonary embolism .

A number of imaging modalities are currently available to evaluate deep venous system in a comprehensive manner allowing correct assessment of presence of thrombosis . Color Doppler ultrasound has become the primary non invasive diagnostic method for DVT.

All patients are going to be examined by color Doppler ultrasound and by direct MDCT venography .

ELIGIBILITY:
Inclusion Criteria:

* female patients in different age groups with gynecological masses detected by clinical examination and different imaging modalities.

Exclusion Criteria:

1. patients with chronic kidney disease in case of contrast .
2. patients complaining from hematological diseases that may cause venous thromboembolism .
3. pregnant patients .
4. patients already diagnosed with deep venous thrombosis.
5. patients not fit for surgery.

Sex: Female
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — female patients in different age groups with gynecological masses detected by clinical examination and different imaging modalities.
Study Population: patients admitted to Assiut University hospitals
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2017-09 (Estimated); Primary Completion 2020-09 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
detection of asymptomatic venous thrombosis | one week before operation
  silent venous thrombosis in gynecological patients with pelvic masses

REFERENCES:
- [Background] Ikeda M, Kan-no H, Hayashi M, Tsukada H, Shida M, Hirasawa T, Muramatsu T, Ogushi Y, Mikami M. Predicting perioperative venous thromboembolism in Japanese gynecological patients. PLoS One. 2014 Feb 26;9(2):e89206. doi: 10.1371/journal.pone.0089206. eCollection 2014. PMID 24586595
- [Background] Qu H, Li Z, Zhai Z, Liu C, Wang S, Guo S, Zhang Z. Predicting of Venous Thromboembolism for Patients Undergoing Gynecological Surgery. Medicine (Baltimore). 2015 Sep;94(39):e1653. doi: 10.1097/MD.0000000000001653. PMID 26426660
- [Background] Goodman LR, Stein PD, Matta F, Sostman HD, Wakefield TW, Woodard PK, Hull R, Yankelevitz DF, Beemath A. CT venography and compression sonography are diagnostically equivalent: data from PIOPED II. AJR Am J Roentgenol. 2007 Nov;189(5):1071-6. doi: 10.2214/AJR.07.2388. PMID 17954642
- [Background] Kelly J, Rudd A, Lewis RR, Hunt BJ. Screening for subclinical deep-vein thrombosis. QJM. 2001 Oct;94(10):511-9. doi: 10.1093/qjmed/94.10.511. No abstract available. PMID 11588209
- [Background] Satoh T, Oki A, Uno K, Sakurai M, Ochi H, Okada S, Minami R, Matsumoto K, Tanaka YO, Tsunoda H, Homma S, Yoshikawa H. High incidence of silent venous thromboembolism before treatment in ovarian cancer. Br J Cancer. 2007 Oct 22;97(8):1053-7. doi: 10.1038/sj.bjc.6603989. Epub 2007 Sep 25. PMID 17895896